CLINICAL TRIAL: NCT06912633
Title: A Randomized, Masked, Sham-Controlled Phase 2 Trial of the Safety of a Single Intravitreal Injection of jCell (Famzeretcel) for the Treatment of Retinitis Pigmentosa (RP)
Brief Title: Safety of a Single, Intravitreal Injection of 6.0M jCell (Famzeretcel) in Retinitis Pigmentosa (RP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: jCyte, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JC02-88
Record Dates: First submitted 2025-03-26; First posted 2025-04-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects, their family members, and clinical staff performing efficacy assessments will be masked to the randomization assignment of subjects. Due to the nature of some safety assessments and the sham treatment, not all study personnel can be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 6.0M jCell injection (Experimental): Single intravitreal injection of 6.0 million retinal progenitor cells into the study eye
  Interventions: Biological: human retinal progenitor cells
- Sham-treated control (Sham Comparator): A mock injection will be performed on the study eye in each control subject
  Interventions: Other: Mock injection

INTERVENTIONS:
Biological: human retinal progenitor cells — Single intravitreal injection of 6.0 million retinal progenitor cells (RPCs)
  Other Names: jCell; famzeretcel
  Arms: 6.0M jCell injection
Other: Mock injection — Pressing the hub of a syringe with no needle against the eye to mimic intravitreal injection. Subjects randomized to the sham control group will undergo identical preparation as the active treatment group immediately prior to treatment, including application of anesthetics.
  Arms: Sham-treated control

SUMMARY:
This study evaluates the safety of a single injection of jCell (famzeretcel) comprising 6.0 million (6.0M) retinal progenitor cells over a six-month study period in a cohort of adult subjects with RP. Additionally, changes in visual function will be evaluated at six months between the active treatment group (6.0M jCell) compared to sham-treated controls.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of RP supported by at least 2 of the following clinical findings: (1) Loss of peripheral vision on formal visual field testing, (2) Symptoms of night blindness or difficulty adjusting to dim light, or (3) Optical coherence tomography (OCT) outer retinal atrophy consistent with RP.
2. Electroretinography (ERG) results that support diagnosis of RP including nondetectable or severely reduced rod responses (defined as less than 30% of the lower limit of normative values for the ERG lab performing the test), with prolonged implicit time OU (i.e., ensure bilateral involvement) and greater rod than cone loss. If genotyping results from a certified genetic testing lab document mutations clearly diagnostic of RP, with no other potential diagnosis of a disease(s) distinct from RP, the genetic test may be used in lieu of an ERG.
3. Subject age ≥ 18 years and ≤ 60 years at time of signing of consent.
4. Interocular BCVA disparity ≤ 15 letters.
5. Central subfield thickness (CST) ≥ 130 µm in the study eye.
6. BCVA no better than 55 letters and no worse than 1 letter using the Early Treatment Diabetic Retinopathy Study (ETDRS) testing protocol in the study eye.
7. Ability to reliably fixate with the study eye at least 75% of the time as indicated by a fixation score of four (4) or five (5) on semi-automated kinetic visual fields.
8. Ability to record at least two reliable trials at a minimum baseline contrast sensitivity reading of 1.28 at a minimum of one spatial frequency using the Beethoven system in the study eye.
9. Central island visual field area (central island contiguous to fixation), of ≥ 50.3 deg2 (~ central island visual field diameter ≥ 8°) in the study eye.
10. Willingness of subject to provide informed consent, including acknowledgement that they are able and willing to attend all required study visits, follow study protocol assessment instructions, travel by air if necessary, and provide Health Insurance Portability and Accountability Act (HIPAA) authorization.
11. Willingness of subject to provide a blood sample for human leukocyte antigen (HLA) typing, if not done previously with available results.
12. Willingness of subject to consent to testing for RP gene mutation typing, if not performed previously with available results.
13. Adequate organ function.
14. Negative active infectious disease screen (active infection with Hepatitis B, C, human immunodeficiency virus [HIV]).
15. A female subject of childbearing potential must have a negative pregnancy test (urine human chorionic gonadotropin) at entry (prior to treatment).
16. Women of childbearing potential must agree to use a medically accepted method of contraception for at least 12 months after jCell injection.
17. For male patients whose partners are of child-bearing potential, willingness to use a medically accepted method of contraception.

Exclusion Criteria:

1. Participation in any clinical trial of a drug intervention within the last 6 months, with the exception of a N-acetyl cysteine (NAC) study.
2. History of ocular treatment with any non-approved, experimental, investigational or neuroprotectant therapy (systemic, topical, intravitreal) or device in either eye, including previous jCyte clinical trials. Individuals with a history of NAC treatment may take part in the study following a 7-day washout period (prior to Baseline testing).
3. Subject is currently breast feeding/pumping or is planning to breast feed/pump during the 12 months after study treatment.
4. Subject is pregnant or intends to become pregnant less than 12 months after jCell injection.
5. Known allergy to gentamicin.
6. History of adverse reaction to dimethyl sulfoxide (DMSO).
7. Prior ocular treatment with corticosteroids (systemic, periocular, intracanalicular or intravitreal - in either eye) within six months of study randomization or the anticipated need for the use of these agents to treat a pre-existing ocular condition.
8. Clinical evidence of history of any eye disease or pathology, other than RP, IN EITHER EYE, that is associated with increased risk of pathology developing in the study eye, that could impair visual function, testing procedures, clinical trial endpoint measurements and/or the outcome of the study. Examples include central serous retinopathy, vitreomacular traction, pattern/vitelliform dystrophy
9. Clinical evidence of history of any eye disease or pathology, other than RP, IN THE STUDY EYE, that could potentially impair visual function, testing procedures, clinical trial endpoint measurements and/or the outcome of the study.
10. Concurrent use of any prohibited therapies.
11. History of prior use of the following medications is prohibited if any retinal/retinal pigment epithelium (RPE) abnormalities are noted in the macula on exam or OCT: Hydroxychloroquine or chloroquine (Plaquenil); Pentosan polysulfate sodium [PPS] (Elmiron); and Interferon (Intron A, Roferon-A, IFN-alpha, alpha interferon).
12. Any mental health issue likely to prevent subject from reliably performing study testing and/or examinations including dementia, schizophrenia, bipolar disorders if not reliably controlled on medications, depression if any history of hospitalization or in-patient treatment or if not sufficiently controlled on medications to enable, in the opinion of the investigator, travel to and compliance with study testing requirements over the study period.
13. Uncontrolled blood pressure defined as systolic pressure > 180mmHg and/or diastolic blood pressure > 110mmHg, while subject is at rest.
14. Any chronic systemic disease requiring continuous treatment with systemic steroids or immunosuppressive agents.
15. History of any disease interfering with the participation in the study according to the investigator judgment, including of any type of cancer that is not in remission or considered cured, diabetes mellitus (history of gestational diabetes is acceptable), renal failure, stroke, transient ischemic attack (TIA), any systemic immune condition, any coagulopathy disorder that is not adequately managed/controlled.
16. Current systemic treatment for a confirmed active infection.
17. For male patients whose co-partners are of child-bearing potential, lack of willingness to use a medically accepted method of contraception, not including the rhythm method, for at least 12 months after jCell injection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety of Intravitreal Injection of 6.0M jCell | 6 months
  Assessed by treatment emergent adverse events, immunogenicity and safety visual assessments

SECONDARY OUTCOMES:
BCVA responder rate (≥ 15 letters) | 6 months
  proportion of responders who achieve at least 15 ETDRS letter improvement in best corrected visual acuity (BCVA) from baseline to 6-months post-treatment
BCVA responder rate (≥ 10 letters) | 6 months
  proportion of responders who achieve at least 10 ETDRS letter improvement in best corrected visual acuity (BCVA) from baseline to 6-months post-treatment
Peak contrast sensitivity (CS) responder rate (≥ 0.3 log CS) | 6 months
  proportion of responders who achieve at least a 0.3 log contrast sensitivity (CS) improvement in peak CS from baseline to 6-months post-treatment
Mean change in VA LV VFQ-48 mobility domain test scores | 6 months
  The VA LV VFQ-48 (VFQ) is used to capture changes in patients' self-reporting of their difficulty with reading, mobility and performing other daily living activities affected by visual impairment. There are 4 scales on the VFQ including Visual Information, Reading, Visual Motor, and Mobility. The data shown in this outcome measure is focused on the fourth scale, Mobility, and is measured in units called logits. Higher positive values on the Mobility score represent better function and less impairment, whereas lower or negatives scores represent worse function or more impairment. Change in the Mobility scale on the VFQ is calculated by taking a subject's score at 6 months and subtracting from it the baseline score.
Mean change in VA LV VFQ-48 visual ability (overall) test scores | 6 months
  The VA LV VFQ-48 (VFQ) is used to capture changes in patients' self-reporting of their difficulty with reading, mobility and performing other daily living activities affected by visual impairment. There are 4 scales on the VFQ including Visual Information, Reading, Visual Motor, and Mobility. A fifth value, Visual Ability, is an aggregate score of the 4 scales, measured in units called logits, and is calculated for each person based on item weighting using Raasch analysis. Visual Ability is used broadly to represent changes in subject-reported outcomes from visit to visit. Higher positive values on the Visual Ability score represent better function and less impairment, whereas lower or negatives scores represent worse function or more impairment. Change in the Visual Ability scale on the VFQ is calculated by taking a subject's score at 6 months and subtracting from it the baseline score.
Mean change in central island visual field area | 6 months
  mean change in central island visual field area (visual field that is contiguous to fixation, excluding peripheral islands), as assessed by semi-automated kinetic perimetry, from baseline to 6-months post-treatment
Mean change in EQ-5D-5L test scores | 6 months
  The EQ-5D-5L is a generic measure of health status consisting of two parts. The first part (the descriptive system) assesses health in five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and provides a descriptive profile that can be used to generate a health state profile. Each health state can be assigned a summary index score, ranging from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health). Changes in health state index and EQ VAS scores are calculated by taking a subject's scores at 6 months and subtracting from them the baseline scores.
Mean change in peak contrast sensitivity (CS) | 6 months
  mean change in peak CS from baseline to 6-months post-treatment
Mean change in BCVA | 6 months
  mean change in best corrected visual acuity (BCVA) from baseline to 6-months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry Klassen, MD, PhD, Principal Investigator — jCyte, Inc
Locations (7):
- United States (7):
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Gavin Herbert Eye Institute, UC Irvine, Irvine, California
  - Retina Consultants Medical Group, Sacramento, California
  - Illinois Retina Associates, Oak Park, Illinois
  - Long Island Vitreoretinal Consultants, Westbury, New York
  - Retina Consultants of Texas: Bellaire Retina Center, Bellaire, Texas